CLINICAL TRIAL: NCT02672800
Title: A Psychosocial Intervention for Bereaved Spousal Caregivers of Persons With Dementia: Adapting the "Finding Balance" Tool
Brief Title: A Psychosocial Intervention for Bereaved Spousal Caregivers of Persons With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Shelley Peacock, Assistant Professor, College of Nursing, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 15-313
Record Dates: First submitted 2016-01-28; First posted 2016-02-03 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Dementia; Bereavement
MeSH Terms: conditions — Dementia

ARMS (2):
- Writing intervention (Experimental)
  Interventions: Behavioral: the Reclaiming Yourself tool
- Control (No Intervention)

INTERVENTIONS:
Behavioral: the Reclaiming Yourself tool — This tool is a behavioural writing intervention, intended to facilitate bereavement for spousal caregivers of persons with dementia
  Arms: Writing intervention

SUMMARY:
The purpose of this study is to evaluate the feasibility and acceptability of a writing intervention (Reclaiming Yourself), intended to facilitate bereavement for spousal caregivers whose partners died with dementia.

DETAILED DESCRIPTION:
The current research is part 3 of a multi-phase project, whose purpose was to examine the experience of bereavement for spousal caregivers to persons with dementia. Based on spouses' shared experiences and the input of experts in the field (i.e. bereavement/dementia researchers, health care providers), an existing writing intervention called the Finding Balance tool was adapted from the context of cancer bereavement to that of dementia.

The purpose of this third phase is to test this adapted writing intervention (Reclaiming Yourself) with bereaved spouses of persons with dementia. Participants will be randomly assigned into one of two groups: treatment (who will receive the tool); and control (who will not be offered the tool until a later stage). The feasibility and acceptability of the intervention will be assessed, as well as the degree to which it facilitated participants' bereavement, ability to find balance, and psychological health.

ELIGIBILITY:
Inclusion Criteria:

* bereaved for three months or longer
* were a caregiver for their spouse with advanced dementia
* English speaking
* willing and able to share their bereavement experience

Exclusion Criteria:

* those with other than a spousal relationship to the person with dementia
* spousal caregivers of persons with another terminal disease
* those bereaved less than 3 months
* those unable to provide consent

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-03; Primary Completion 2017-12 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Inventory of Daily Widowed Life (IDWL)- change at 1 and 2 months post-intervention | The measure will be administered pre-intervention, 1 month following the introduction of the intervention, and 2 months following the introduction of the intervention
  Measure of finding balance in bereavement
Center for Epidemiologic Studies Depression Scale- Revised (CESD-R)- change at 1 and 2 months post-intervention | The measure will be administered pre-intervention, 1 month following the introduction of the intervention, and 2 months following the introduction of the intervention
  Measure of depressive symptoms
Texas Revised Inventory of Grief, Present Feelings- change at 1 and 2 months post-intervention | The measure will be administered pre-intervention, 1 month following the introduction of the intervention, and 2 months following the introduction of the intervention
  Measure of grief

SECONDARY OUTCOMES:
Semi-structured qualitative evaluation interviews | Post intervention (after 1 month)
  Measure of the feasibility and acceptability of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Shelley Peacock, RN, PhD, Principal Investigator — University of Saskatchewan
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada